CLINICAL TRIAL: NCT02928458
Title: Clinical and Financial Impact of an Evidenced-Based Adhesive Small Bowel Obstruction Management Protocol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1609-39
Record Dates: First submitted 2016-07-18; First posted 2016-10-10 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Intestinal Obstruction
MeSH Terms: conditions — Intestinal Obstruction | interventions — Iohexol; Diatrizoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omnipaque (Active Comparator): Arm 1
  Interventions: Drug: Omnipaque
- MD-Gastroview (Active Comparator): Arm 2
  Interventions: Drug: MD-Gastroview

INTERVENTIONS:
Drug: Omnipaque
  Arms: Omnipaque
Drug: MD-Gastroview
  Arms: MD-Gastroview

SUMMARY:
This research study is for patients with adhesive small bowel obstruction (ASBO). ASBO is a condition in which the small intestine gets blocked due to scars called adhesions. To see the blockage, a contrast agent is given and an x-ray is taken of the belly (abdomen). MD Gastroview and omnipaque are two contrast agents that may be given as part of your normal care for ASBO. This study hopes to see if one is better than the other.

DETAILED DESCRIPTION:
Small bowel obstruction is a common general surgical diagnosis providing a significant proportion (16%) of the emergency general surgery admissions. Unfortunately, there is a paucity of clear, well defined management protocols for this very common problem which results in a wide array of management techniques used by the general surgeon. It has already been shown that CT scan with IV contrast is the most accurate method of identifying strangulated bowel, a diagnosis that requires urgent surgical intervention(4). There is no variability in this aspect of the treatment arm for ASBO, rather the variability is found in the medical management of ASBO. Nasogastric tube (NGT) decompression is a universal component of non-operative management but the duration of NGT therapy and the definition of failed medical management requiring surgery lack a clear consensus. It is this aspect of the management of ASBO that I am hoping to better define. Water soluble contrast (MD-Gastroview) has been shown to be both diagnostic and therapeutic in the management of ASBO decreasing length of stay in this patient population. Not only does it expedite the resolution of ASBO, but is also yields objective evidence whether or not ASBO will resolve with medical management alone, therefore decreasing delay in the inevitable surgical intervention.

The hypothesis of this study is that the implementation of an evidence based adhesive small bowel obstruction protocol can reduce length of stay and reduce the financial burden on the health care system regarding this common general surgical problem. A second hypothesis is that MD-Gastroview and omnipaque will have similar properties regarding their diagnostic and therapeutic impact on ASBO.

ELIGIBILITY:
Inclusion Criteria:

* Principle diagnosis of adhesive small bowel obstruction

Exclusion Criteria:

* Evidence of strangulation on initial CT scan leading to emergent operation
* Any known allergy to either contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Compare average length of stay for patients admitted with ASBO prior to and after implementation of this protocol. | Three years

SECONDARY OUTCOMES:
Compare statistically significant results relating to differences in the diagnostic and therapeutic effects of MD-Gastroview and omnipaque. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Behm, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- The Guthrie Clinic, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No